CLINICAL TRIAL: NCT00901160
Title: Pilot Study for the Prediction of Post-operative Thrombotic and Bleeding Complications in Non-cardiac Surgery Using Thromboelastography (TEG®) and Platelet Mapping Assay (PMA™) in Patients on Anti-platelet Agents
Brief Title: Thromboelastography (TEG®) and Platelet Function in Patients on Anti-platelet Agents
Status: Terminated | Type: Observational
Why Stopped: Unable to get funding
Sponsor: McMaster University (Other)
Collaborators: University Health Network, Toronto (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 07-468
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Blood Clotting
Keywords: thromboelastography; post-operative complications; anti-platelet agents; prospective; pilot; patients taking anti-platelet agents
MeSH Terms: conditions — Thrombosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical patients: Blood will be taken from patients who are on anti-platelet medication and are having surgery that requires an overnight stay. This is a pilot study to see if Thromboelastography® and Platelet Mapping Assay™ will be able to predict if a patient is at risk for a bleeding or a clotting problem after surgery.
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: blood test — Blood will be taken from patients shortly after surgery in the recovery room in order to perform Thromboelastography® and Platelet Mapping Assay™ tests.

SUMMARY:
Can a post-operative analysis using a simple blood test (Thromboelastography(TEG®)) and Platelet Mapping Assay (PMA™) be able to detect the occurence of clotting or bleeding complications in patients on blood thinning (anti-platelet) agents?

DETAILED DESCRIPTION:
Two hundred patients coming for surgery who are taking anti-platelet medications will be enrolled in this study as a pilot, to determine the feasibility for a larger study. A simple blood test for clotting function will be done after surgery. Patients will be assessed daily during their hospital stay to determine if they have any clotting or bleeding complications. For analysis, groups will be divided into normal and increased or decreased ability to make a blood clot based on the TEG® and PMA™ test done. Complications will be recorded for each group and analyzed to determine if there is any difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* patients on aspirin and/or clopidogrel for at least 10 days, having non-ambulatory, non-cardiac, elective surgery

Exclusion Criteria:

* anemia (Hb < 100) or thrombocytopenia (platelet count < 80), having any known clotting abnormalities
* family history of clotting abnormalities
* concurrently on NSAIDs, warfarin therapy or other treatments affecting platelet function
* renal impairment (Cr > 110 mg for females or Cr > 125 mg) or INR > 1.2

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are having non-ambulatory, non-cardiac, elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Patients undergoing non-cardiac (non-ambulatory) surgery and are on anti-platelet agents, is hyper or hypocoagulability based on TEG® and PMA™ associated with increased risk of thrombotic and bleeding complications. | 1 month

SECONDARY OUTCOMES:
Is hypercoagulability based on TEG®(MA) and PMA™ associated with increased risk of the following events post-op: MI, stroke, PE, DVT, death? | 1 month
Is hypo-coagulation status associated with lower levels of nadir and discharge hemoglobin/hematocrit and increased transfusion? | 1 month
Is coagulation status associated with hospital length of stay? | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Summer Syed, M.D., Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network, Toronto, Ontario